CLINICAL TRIAL: NCT06541145
Title: Impact of Bacterial Decolonization on Bacterial Burden Within Maternal-infant Dyads
Brief Title: Bacterial Decolonization Within Dyads
Acronym: BADMC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00115222
Record Dates: First submitted 2024-08-02; First posted 2024-08-07 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Bacterial Colonization
Keywords: Maternal; Infant; Neonatal; Resistant; Antimicrobial
MeSH Terms: interventions — Mupirocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Maternal Skin Decolonization (Experimental): These decolonization methods have been safely tolerated in adults and children. We propose a combination of intranasal mupirocin and chlorhexidine baths for a 5-day decolonization regimen targeting pregnant women in their third trimester prior to delivery
  Interventions: Drug: Mupirocin; Drug: Chlorhexidine baths
- Baseline or control dyads (No Intervention): Maternal-infant dyads without exposure to skin decolonization treatment

INTERVENTIONS:
Drug: Mupirocin — Participants will place a pea-sized amount (or approximately 1cm ribbon) of 2% mupirocin ointment (Duke formulary) on a cotton swab and gently massage it into the anterior nares twice daily for 5 days.
  Other Names: Bactroban
  Arms: Maternal Skin Decolonization
Drug: Chlorhexidine baths — Participants will be instructed to use pre-packaged chlorhexidine cloths. Each cloth will be used to wipe designated body areas (i.e., arms, legs, chest and neck, back and perineum) once a day for 5 days. These are inexpensive cloths that are easy to use and have been shown to be effective at eradicating Staph aureus carriage. Ideally, participants will be instructed not to rinse off immediately after using the cloths. Baths should be performed on the same 5 days as they apply the intranasal mupirocin.
  Other Names: CHG cloths
  Arms: Maternal Skin Decolonization

SUMMARY:
The goal of this study is to measure bacterial burden, specifically Staph aureus, and how it spreads between mothers and their infants. Researchers will evaluate if the amount of bacteria on their skin remains the same after mothers use a skin antisepsis treatment prior to delivering their infants. The investigators also aim to assess participant interest in and compliance with skin antisepsis treatments. The hypothesis is that increased maternal interest will align with increased treatment compliance.

DETAILED DESCRIPTION:
Few studies have assessed the clinical epidemiology of bacterial transmission among mother-infant dyads in hospitalized and community settings. In an era of rising antimicrobial resistance, the epidemiology of colonization and infections are also changing. Maternal factors account for infants' early exposure to bacteria. Maternal colonization with multi-drug resistant (MDR) bacteria portends a high likelihood of transmission to the infant.

As methicillin resistant Staph aureus (S. aureus) bacteria remain among the top causes of pediatric infections, the presence of these species among mothers and infants can be used to assess antimicrobial resistance, colonization and transmission in maternal-infant dyads. S. aureus is a uniquely interesting pathogen in the perinatal period. MRSA nasal colonization is a sensitive predictor of bloodstream, genitourinary and respiratory infections. Also, parental colonization with S. aureus is typically concordant with infants' colonizing and infecting S. aureus strains. In tandem, there have been numerous studies assessing the utility and impact of MRSA decolonization for high risk patients. This project creates a unique opportunity for in-depth microbiological analyses of maternal-infant dyads.

Design & Procedures: S. aureus skin decolonization methods have been safely tolerated in adults and children. The investigators propose a combination of intranasal mupirocin and chlorhexidine baths for a 5-day decolonization treatment targeting pregnant women already consented to participate in a longitudinal cohort - Project HOPE cohort. The investigators will aim for maternal participation in their third trimester. The decolonization regimen will include:

1. Intranasal mupirocin - Participants will place a pea-sized amount (or approximately 1cm ribbon) of 2% mupirocin ointment on a cotton swab and gently massage it into the anterior nares twice daily for 5 days.
2. Chlorhexidine baths - Participants will be instructed to use pre-packaged chlorhexidine cloths. Each cloth will be used to wipe designated body areas (i.e., arms, legs, chest and neck, back and perineum) once a day for 5 days. These are inexpensive cloths that are easy to use and have been shown to be effective at eradicating Staph aureus carriage. Ideally, participants will be instructed not to rinse off immediately after using the cloths. Baths should be performed on the same 5 days as they apply the intranasal mupirocin.

Evaluation of decolonization protocol compliance: The investigators will provide verbal and printed instructions in participants' preferred languages (English or Spanish). The research team will conduct two weekly check-ins - one during the treatment week and the other during the subsequent week. The investigators will also conduct online surveys to gauge decolonization tolerance and self-reported completion rates. When plausible, participants will be asked to return the mupirocin tube at their next routinely scheduled visit to confirm appropriate use.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be enrolled in longitudinal study Project HOPE1000.

Exclusion Criteria:

* Participants not enrolled in Project HOPE1000 will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-21 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Staph aureus burden within maternal-infant dyads after exposure to a decolonization regimen | 12 months
  Mucosal swabs collected in the parent study, Project HOPE biorepository are stored in RNALater to assess burden by PCR (polymerase chain reaction) at a later date.
Staph aureus epidemiology within maternal-infant dyads after exposure to a decolonization regimen | 12 months
  S. aureus isolates will undergo spa typing for comparison.
Participant interest in skin decolonization | 12 months
  Measured by a descriptive survey, Perception of Safety Survey for Pregnant Women Undergoing Skin Treatment.
Participant compliance with skin decolonization | 12 months
  Measured by a descriptive survey, Perception of Safety Survey for Pregnant Women Undergoing Skin Treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ibukunoluwa Kalu, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No